CLINICAL TRIAL: NCT06174272
Title: Transitional Care Program vs Standard of Care in Cirrhosis With Volume Overload: A Pilot Study
Brief Title: Transitional Care Program for Fluid Overload in Cirrhosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Karen Krok, Professor of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00023071
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis, Liver
Keywords: ascites; anasarca; edema
MeSH Terms: conditions — Liver Cirrhosis; Ascites; Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transitional Care Program (Experimental): Participants will receive a digital scale and monitoring log, educational material, a phone call within 72 hours of discharge and weekly for 8 weeks, and a follow up appointment with a hepatologist within 4 weeks of discharge.
  Interventions: Behavioral: Transitional Care Program
- Standard of Care (No Intervention): Participants will be given typical discharge and follow up instructions.

INTERVENTIONS:
Behavioral: Transitional Care Program — Intensive monitoring post discharge for cirrhosis and fluid overload
  Arms: Transitional Care Program

SUMMARY:
The goal of this clinical trial is to learn about an intensive monitoring plan (transitional care program) in patients with cirrhosis and excessive swelling that are going to be discharged from the hospital.

The main question[s] it aims to answer are:

* How much time and what resources are needed to run such a program
* How well do patients follow up with the phone calls, bloodwork, and doctor appointments?
* Do the patients enrolled in the program have less need for hospitalization later, less kidney injury, better fluid control, and/or better survival compared to patients that are not in the program?

Participants will

* Be given a digital scale and a binder with educational material and a log to monitor their weights after discharge from the hospital
* Receive a phone call from the study team within 72 hours of discharge and weekly
* Be given a follow up appointment with hepatology within 4 weeks of discharge

Researchers will compare participants in this program to patients that receive normal care to see if there are differences in need for hospitalization later, kidney injury, fluid control, and/or survival.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years of age.
* Inpatient at Penn State Health, Milton S. Hershey Medical Center.
* Diagnosis of cirrhosis.
* Hospitalized with fluid overload (ascites and/or significant anasarca/edema) requiring diuretic therapy.
* English speaking

Exclusion Criteria:

* Placement of a TIPS.
* Ascites from an etiology other than cirrhosis, such as malignancy, heart failure, pancreatitis, nephrotic syndrome.
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
feasibility of the program | all 8 weeks of each participant
  how much time does it take to review material and complete phone calls
Number of instances of weight monitoring | 8 weeks for each participant
  at home monitoring weight
Number of successful phone calls | 8 weeks for each participant
  weekly phone call with participant
Number of follow up visits | 8 weeks for each participant
  lab visits, primary care visits, hepatology visits

SECONDARY OUTCOMES:
Number of Hospitalizations per participant | 12 months
  number of admissions to the hospital
Number of subjects that develop Acute Kidney Injury | 12 months
  Creatinine increase of >0.3g/dL
Number of subjects that continue to have volume overload | 12 months
  persistent weight above dry weight and/or ongoing ascites/lower extremity edema/pleural effusion
Number of subjects that expire | 12 months
  subject death

CONTACTS AND LOCATIONS:
Overall Officials: Karen L Krok, MD, Principal Investigator — Penn State College of Medicine
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No